CLINICAL TRIAL: NCT01802775
Title: A Randomized, Open-Label, Parallel-Group, Multi-Center Study Of Adding Edoxaban Or Clopidogrel To Aspirin To Maintain Patency In Subjects With Peripheral Arterial Disease Following Femoropopliteal Endovascular Intervention
Brief Title: Edoxaban in Peripheral Arterial Disease
Acronym: ePAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DU176b-E-U210; 2012-003009-88 (EudraCT Number)
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — edoxaban; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- edoxaban/aspirin (Experimental): Open label edoxaban will be provided. Subjects randomized to this treatment arm will receive edoxaban 60 mg once daily (QD) (two 30 mg tablets) for a total of approximately 3 months on a background of aspirin 100 mg QD.
  Interventions: Drug: edoxaban; Drug: Aspirin
- clopidogrel/aspirin (Active Comparator): Open label clopidogrel will be provided. Subjects randomized to this treatment arm will receive clopidogrel 75 mg QD (one 75 mg tablet) for a total of approximately 3 months on a background of aspirin 100 mg QD. A loading dose of clopidogrel 300 mg (four 75mg tablets) will be given to subjects as the first dose as early as possible after adequate hemostasis (i.e., within 4 hours of hemostasis).
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: edoxaban
  Arms: edoxaban/aspirin
Drug: Clopidogrel — 75mg tablet
  Other Names: Plavix
  Arms: clopidogrel/aspirin
Drug: Aspirin

SUMMARY:
This study is a randomized, open-label, blinded endpoint, parallel-group, active-control, multi-center, proof-of-concept study in subjects with Peripheral Arterial Disease (PAD), designed to assess the safety and potential efficacy of adding edoxaban to aspirin following femoropopliteal endovascular intervention, with or without stent placement, relative to current treatment practice with clopidogrel and aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects older than the minimum legal adult age (country specific);
* Rutherford stages 2-5 provided there are no ulcerations on the heel and/or exposed tendon and/or bone;
* Superficial femoral above knee-popliteal ( 3 cm proximal to the medial femoral condyle) lesion and ≥ 50% stenosis or occlusion;
* At least one run-off vessel to the foot with or without additional endovascular intervention;
* Successful intervention, defined as angiographic confirmation of ≤ 30% residual stenosis and absence of flow limiting dissection;
* Adequate hemostasis at the vascular access site within 24 hours of intervention;
* A subject is also eligible if they have undergone additional successful endovascular intervention(s) during the index intervention;
* Able to provide signed informed consent.

Exclusion Criteria:

* Calculated Creatinine Clearance < 30 ml/min;
* Femoral or popliteal aneurysm;
* Adjunctive use of thrombolytics;
* Any extravasation or distal embolization not successfully treated;
* Uncontrolled hypertension as judged by the investigator (e.g., systolic blood pressure > 170 mmHg or diastolic blood pressure > 100 mmHg despite antihypertensives);
* Aspirin intolerance;
* Clopidogrel intolerance;
* Contraindication for anticoagulants or antiplatelets and any other contraindication listed in the local labeling of aspirin and/or clopidogrel;
* Active bleeding or known high risk for bleeding or history of intracranial, or spontaneous intraocular, spinal retroperitoneal or intra-articular bleeding; overt gastrointestinal (GI) bleeding or active ulcer within the previous year;
* Subjects receiving dual antiplatelet or anticoagulant therapy at the time of randomization; subjects receiving pre-interventional loading dose of clopidogrel or other P2Y12 receptor antagonists;
* Treatment with cilostazol within 24 hours of randomization;
* Subjects receiving prohibited concomitant medications [fibrinolytics, chronic use of non steroidal anti-inflammatory drugs (NSAIDS) > 4 days per week, and oral or parenteral non-aspirin NSAIDs and strong P-gp inhibitors];
* Prior stroke or myocardial infarction (MI) or acute coronary syndrome within 3 months;
* Chronic liver disease [alanine transaminase (ALT) and/or aspartate transaminase (AST) ≥ 2 × upper limit of normal; total bilirubin (TBL) ≥ 1.5 × upper limit of normal]; however, subjects whose elevated TBL is due to known Gilbert"s syndrome may be included in the study;
* Prior history of a positive test for Hepatitis B antigen or Hepatitis C antibody;
* Subjects who received any investigational drug or device within 30 days prior to randomization, or plan to receive such investigational therapy during the study period;
* Subjects previously randomized to an edoxaban (DU-176b) study;
* Women of childbearing potential without proper contraceptive measures (i.e. a method of contraception with a failure rate < 1 % during the course of the study including the observational period) and women who are pregnant or breast feeding;
* Subjects with the following diagnoses or situations:

Active malignancy except for adequately treated non-melanoma skin cancer or other non-invasive or in-situ neoplasm (e.g., cervical cancer in situ); Concurrent treatment with cancer therapy (drugs, radiation, and/or surgery); Other significant active concurrent medical illness or infection; Life expectancy < 12 months;

* Subjects who are unlikely to comply with the protocol (e.g., uncooperative attitude, inability to return for subsequent visits, and/or otherwise considered by the Investigator to be unlikely to complete the study);
* Subjects with any condition that, in the opinion of the Investigator, would place the subject at increased risk of harm if he/she participated in the study;
* History of heparin-induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2013-02-06 (Actual); Primary Completion 2014-12-03 (Actual); Study Completion 2014-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (42):
- United States (26):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Beverly Hills, California
  - Los Angeles, California
  - Orange, California
  - New Haven, Connecticut
  - Hollywood, Florida
  - Jacksonville, Florida
  - Aurora, Illinois
  - Iowa City, Iowa
  - New Orleans, Louisiana
  - Lewiston, Maine
  - Boston, Massachusetts
  - Flint, Michigan
  - Ypsilanti, Michigan
  - Teaneck, New Jersey
  - New York, New York
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Camp Hill, Pennsylvania
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Austin, Texas
  - San Antonio, Texas
- Austria (3):
  - Graz
  - Innsbruck
  - Vienna
- Belgium (3):
  - Edgem, Edegem
  - Ghent
  - Leuven
- Germany (2):
  - Bad Krozingen
  - Leipzig
- Israel (4):
  - Afula
  - Jerusalem
  - Tel Aviv
  - Tel Litwinsky
- Netherlands (2):
  - Rotterdam
  - Utrecht
- Switzerland (2):
  - Bern
  - Zurich

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Moll F, Baumgartner I, Jaff M, Nwachuku C, Tangelder M, Ansel G, Adams G, Zeller T, Rundback J, Grosso M, Lin M, Mercur MF, Minar E; ePAD Investigators. Edoxaban Plus Aspirin vs Dual Antiplatelet Therapy in Endovascular Treatment of Patients With Peripheral Artery Disease: Results of the ePAD Trial. J Endovasc Ther. 2018 Apr;25(2):158-168. doi: 10.1177/1526602818760488. PMID 29552984
- [Derived] Tangelder MJ, Nwachuku CE, Jaff M, Baumgartner I, Duggal A, Adams G, Ansel G, Grosso M, Mercuri M, Shi M, Minar E, Moll FL. A review of antithrombotic therapy and the rationale and design of the randomized edoxaban in patients with peripheral artery disease (ePAD) trial adding edoxaban or clopidogrel to aspirin after femoropopliteal endovascular intervention. J Endovasc Ther. 2015 Apr;22(2):261-8. doi: 10.1177/1526602815574687. PMID 25809373

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 275 subjects were screened, of these 203 subjects were randomized into the study, with 101 subjects in the edoxaban group and 102 subjects in the clopidogrel group.
Groups:
- Clopidogrel: Open-label clopidogrel with aspirin
- Edoxaban: Open-label edoxaban with aspirin
Period: Overall Study
Arm/Group | Clopidogrel | Edoxaban
Started | 102 | 101
Received Drug (Safety Analysis Set) | 101 | 100
Completed | 96 | 89
Not Completed | 6 | 12
Not completed — Death | 0 | 3
Not completed — Reason not provided | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intention to treat - all participants enrolled in the trial
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel | Edoxaban | Total
Number analyzed (Participants) | 102 | 101 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.55) | 68 (10.36) | 67.4 (9.49)
Age, Customized [Count of Participants; unit: Participants]
  Adults 18-64 years of age | 33 | 30 | 63
  From 65 to 84 years of age | 68 | 65 | 133
  85 years of age and over | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 34 | 58
  Male | 78 | 67 | 145
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 13 | 15 | 28
  Netherlands | 5 | 8 | 13
  Belgium | 6 | 9 | 15
  United States | 47 | 42 | 89
  Israel | 7 | 5 | 12
  Switzerland | 13 | 12 | 25
  Germany | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Relevant Bleeding During Treatment
Description: Percentage of participants with clinically relevant bleeding, defined as major bleeding or clinical relevant non-major bleeding, in the on-treatment period based on International Society of Thrombosis and Haemostasis (ISTH)
Time Frame: at 3 months
Population: Safety Analysis Set, defined as all participants who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clopidogrel | Edoxaban
Number analyzed (Participants) | 101 | 100
percentage of participants
  Including Access Site Bleeding (IASB) | 8 [3.5 to 15.0] | 11 [5.6 to 18.8]
  Excluding Access Site Bleed (EASB) | 6 [2.2 to 12.5] | 6 [2.2 to 12.6]

2. Primary Outcome: Percentage of Participants With First Re-stenosis / Re-occlusion
Description: Percentage of participants with re-stenosis/re-occlusion during treatment within 6 months - only the first occurrence of re-stenosis / re-occlusion was counted for each participant
Time Frame: within 6 months
Population: Modified Intent-to-Treat (mITT), defined as all randomized subjects who received at least one dose of the study study and had at least one post-dose duplex scanning
Measure: Number; unit: percentage of participants
Arm/Group | Clopidogrel | Edoxaban
Number analyzed (Participants) | 95 | 94
percentage of participants | 34.7 | 30.9
Statistical Analysis 1: Comparison: Clopidogrel vs Edoxaban; Treatment difference was edoxaban - clopidogrel. For the treatment difference, 95% Confidence interval was calculated using a normal approximation to the binomial distribution; Test type: Other; Treatment Difference = -3.9, 95% CI 2-sided [-17.3 to 9.5]

3. Secondary Outcome: Percentage of Participants With Major, Clinically Relevant Non-major (CRNM), and Minor Bleeding During Treatment
Description: The percentage of participants with major, clinically relevant non-major, and minor bleeding occurring during treatment, within 3 months
Time Frame: within 3 months
Population: Safety Analysis Set, defined as all participants who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clopidogrel | Edoxaban
Number analyzed (Participants) | 101 | 100
percentage of participants
  IASB : Major Bleeding | 5 [1.6 to 11.2] | 1 [0 to 5.4]
  IASB: CRNM Bleeding | 4 [1.1 to 9.8] | 10 [4.9 to 17.6]
  IASB: Minor Bleeding | 20.8 [13.4 to 30] | 20 [12.7 to 29.2]
  EASB : Major Bleeding | 4 [1.1 to 9.8] | 1 [0 to 5.4]
  EASB : CRNM Bleeding | 3 [0.6 to 8.4] | 5 [1.6 to 11.3]
  EASB : Minor Bleeding | 17.8 [10.9 to 26.7] | 19 [11.8 to 28.1]

4. Secondary Outcome: Safety Assessments
Description: Number of participants with serious adverse events (SAEs) within 6 months
  Note: Based on changes to the database structure, clinically significant changes in physical or laboratory parameters are recorded as adverse events (AEs). Details of non-serious adverse events are reported at the 5% reporting threshold in the AE module, as is all-cause mortality.
Time Frame: within 6 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Edoxaban
Number analyzed (Participants) | 101 | 100
Participants | 30 | 31

5. Secondary Outcome: Number of Adjudicated Major Adverse Cardiovascular Events During the Overall Study Period
Description: Number of Adjudicated Major Adverse Cardiovascular Events (MACE) which is a composite of non-fatal myocardial infarction (MI), non-fatal stroke and cardiovascular death
Time Frame: within 6 months
Population: mITT Set 1 (Safety Analysis Set), defined as the participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Edoxaban
Number analyzed (Participants) | 101 | 100
Participants | 1 | 3

6. Secondary Outcome: Number of Participants With Amputations
Description: Number of participants with amputations within 6 months
Time Frame: within 6 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Edoxaban
Number analyzed (Participants) | 101 | 100
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: From the first dose to the end of the study (6 months)
Arm/Group | Clopidogrel | Edoxaban
All-Cause Mortality (participants affected / at risk) | 0/101 | 3/100
Serious Adverse Events (participants affected / at risk) | 30/101 | 31/100
Other Adverse Events (participants affected / at risk) | 23/101 | 32/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clopidogrel (N=101) | Edoxaban (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 2
ANGINA PECTORIS (Cardiac disorders) | 1 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
BRADYCARDIA (Cardiac disorders) | 1 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 2
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 0
CHEST PAIN (General disorders) | 2 | 2
NECROSIS (General disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 1
CLOSTRIDIUM COLITIS (Infections and infestations) | 1 | 0
GANGRENE (Infections and infestations) | 1 | 2
INFECTED SKIN ULCER (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
UROSEPSIS (Infections and infestations) | 1 | 0
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1 | 3
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 | 4
WOUND (Injury, poisoning and procedural complications) | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 0
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 0
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 1 | 0
ALCOHOL ABUSE (Psychiatric disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 1
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 0 | 2
HAEMORRHAGE (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
INTERMITTENT CLAUDICATION (Vascular disorders) | 4 | 2
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 3 | 1
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 2 | 2
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 2 | 3
PERIPHERAL EMBOLISM (Vascular disorders) | 1 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clopidogrel (N=101) | Edoxaban (N=100)
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 | 6
Creatinine renal clearance decreased (Investigations) | 3 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Dizziness (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A study site may not publish results of a study until after a coordinated multicenter publication has been submitted for publication or until one year after the study has ended, whichever occurs first. The site may publish the results with proper regard to the protection of subjects' identities, provided that sponsor (including legal and intellectual property) has had the opportunity to review and comment on the proposed publication prior to its being submitted for publication.